CLINICAL TRIAL: NCT01590511
Title: Echocardiographic Prediction of Fluid Responsiveness After a Mini-fluid Challenge in Non-ventilated Patients With Shock
Acronym: IVT NonVent
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2012/XB-02; 2012-A00500-43 (Other: RCB number)
Record Dates: First submitted 2012-04-30; First posted 2012-05-03 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-12

CONDITIONS: Shock; Circulatory Failure
Keywords: mini fluid challenge; subaortic velocity time integral
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- The study population: Patients in the emergency room or intensive care in acute circulatory failure without ventilatory support.

SUMMARY:
The main objective of this study is to show that the variation of the subaortic velocity time integral after a mini test by filling 100 cc of normal saline over 1 minute (ΔITV100) is predictive of response to filling (defined as an increase in aortic velocity time integral measured by transthoracic ultrasound over 15% after administration of 500 cc of normal saline over 15 minutes) in non-ventilated shock patients.

DETAILED DESCRIPTION:
The secondary objectives of this study include:

* To determine the sensitivity and specificity of the variation of the velocity time integral after administration of 100 cc of normal saline over 1 minute (ΔITV100) to predict the response to the filling.
* To study the inter-observer variation of ΔITV100 measurement.
* To compare ΔITV100 to other clinical and radiological parameters for predicting response to filling (initial value of the subaortic velocity time integral, variation in mitral E wave, E / A, respiratory variation of the diameter of the inferior vena cava, marbling clinical evolution score.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* Systolic blood pressure (SBP) < 90 mmHg
* Signs of inadequate cardiac output: urine output <0.5 ml / kg / h for more than two hours, hyperlactataemia
* Requires amines to maintain an SBP ≥ 90 mmHg or inability to lower amines or requires an increase in amines

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient (or his/her person-of-trust) refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant, parturient, or breastfeeding
* The patients has a contraindication for a treatment necessary for this study
* Cardiogenic shock
* Acute pulmonary edema
* Moribund patient
* Non echogenic patient
* Patient with cardiac arrhythmia
* Patients for whom the passive leg raising test is contraindicated (hyper intra-abdominal pressure, pelvic or lower limb trauma)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the emergency room or intensive care in acute circulatory failure without ventilatory support.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2013-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in the subaortic velocity time integral after 100cc of normal saline over 15 minutes (cm^2) | baseline; 26 minutes

SECONDARY OUTCOMES:
Change if the subaortic velocity time integral after a passive leg raising trial (cm^2) | baseline; 15 minutes
Change in heart rate after the "mini-fluid challenge" | baseline; 26 minutes
  (bpm,%)
Change in mean arterial pressure after the "mini-fluid challenge" (mmHg) | baseline; 26 minutes
Change in mitral E wave (cm / s) after the "mini-fluid challenge" | baseline; 26 minutes
Change in the E/A ratio after the "mini-fluid challenge" | baseline; 26 minutes
Change in the Marbrure clinical score after the "mini-fluid challenge" | baseline; 26 minutes
Change in lower vena cava diameter | baseline; 8 minutes
  (DiameterMax-DiameterMin) / DiameterMax (cm;%)

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Bobbia, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France